CLINICAL TRIAL: NCT02425800
Title: Optimizing Human Prostate Extracellular Matrix as a Structure for Maintenance and Studying of Prostate Cancer Stem Cells
Brief Title: Human Prostate Tissue Model to Maintain and Study Prostate Cancer Stem Cells
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00031636; NCI-2015-00377 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 85A15 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2015-03-24; First posted 2015-04-24 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Benign Prostatic Hyperplasia; Prostate Carcinoma
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — prostate tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (human prostate tissue model): Tissue samples are collected from patients with benign prostatic hyperplasia for decellularization and preparation as human extracellular matrix for growing human prostate CSCs. Tissue samples are also collected from patients with prostate cancer for the analysis of TROP2+ cells by flow cytometry. Cytology Specimen Collection Procedure. Laboratory Biomarker Analysis.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of tissue samples
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This pilot research trial studies the use of a human prostate tissue model to maintain and study prostate cancer stem cells. A human prostate tissue model uses leftover tissue that was removed during surgery from patients with non-cancerous enlargement of the prostate (benign prostatic hyperplasia) and may create an environment similar to the natural environment of the human body. Prostate cancer stem cells are cells that cause cancer to grow. Using real tissue to create an environment to study stem cells may help doctors learn more about how they work and how they respond to treatments.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To optimize a decellularized prostate tissue model for the maintenance of prostate cancer stem cells.

SECONDARY OBJECTIVES:

I. To investigate the self-renewal and differentiation ability of human prostate cancer stem cells (CSCs) (tumor-associated calcium signal transducer 2 [TROP2]+ cells) in the above mentioned decellularized prostate tissue model.

II. To compare the number of CSCs according to key patient characteristics, including race, age, Gleason, metastasis status, and previous cancer treatment(s).

OUTLINE:

Tissue samples are collected from patients with benign prostatic hyperplasia for decellularization and preparation as human extracellular matrix for growing human prostate CSCs. Tissue samples are also collected from patients with prostate cancer for the analysis of TROP2+ cells by flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

* Male patients scheduled for a prostatectomy
* Ability to understand and the willingness to sign an Institutional Review Board (IRB)-approved informed consent document

Exclusion Criteria:

* Patients with prostate involvement secondary and as a result of metastasis or spread of cancerous cells from other organs

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men scheduled for a prostatectomy
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-07-28 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Percent of viable injected cells | Up to 4 weeks
  Optimization of a decellularized prostate tissue model for the maintenance of prostate cancer stem cells, as measured by the viability of the injected cells at different time points (1 day, 2 days, 3 days, 1 week, 2 weeks, 3 weeks, and 4 weeks) will be evaluated. For each day the percent viable and associated confidence interval will be reported.
Ability to make spheres (cluster of cells) | Up to 1 year
  Also to evaluate the primary objective it will be determined if cells are able to make spheres and if so, confidence intervals for the proportion of injected cells that are able to make spheres will be estimated and provided.
Ratio of spheres to the amount of injected cells | Up to 1 year
  Also to evaluate the primary objective it will be determined if cells are able to make spheres and if so, confidence intervals for the proportion of injected cells that are able to make spheres will be estimated and provided.

SECONDARY OUTCOMES:
Number of alive cells (using flow cytometry) | Up to 28 days
  To address the secondary objective of investigating the self-renewal and differentiation ability of human prostate CSCs (TROP2+ cells) decellularized prostate tissue model, the number of alive cells will be observed and an estimate (with confidence interval) of the percentage of the TROP2 positive cells will be obtained at days 3, 7, 14, 21, and 28.
Percentage of the TROP2 positive cells (using flow cytometry) | Up to 28 days
  To address the secondary objective of investigating the self-renewal and differentiation ability of human prostate CSCs (TROP2+ cells) decellularized prostate tissue model, the number of alive cells will be observed and an estimate (with confidence interval) of the percentage of the TROP2 positive cells will be obtained at days 3, 7, 14, 21, and 28.
Ability of cells to make glandular structures by observing the structure under microscope and performing immunostaining for epithelial markers like E-Cadherin, beta-catenin | Up to 1 year
  Estimates and confidence intervals for the percent of cells that are able to make glandular structures will also be provided.
Number of CSCs | Up to 1 year
  The relationships between patient characteristics (including race, age, Gleason, metastasis status, and previous cancer treatment[s]) and the number of CSC's will also be investigated. An estimate of the number of CSC's for each level of categorical characteristics and a correlation for those patient characteristics which are continuous will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Ashok K Hemal, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina